CLINICAL TRIAL: NCT00005205
Title: Incidence of Diabetes and Cardiovascular Disease in Mexican Americans
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1084; R01HL036820 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Myocardial Infarction; Angina Pectoris; Death, Sudden, Cardiac; Cerebrovascular Disorders; Peripheral Vascular Diseases; Coronary Disease; Diabetes Mellitus, Non-insulin Dependent; Diabetes Mellitus
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Myocardial Infarction; Angina Pectoris; Death, Sudden, Cardiac; Cerebrovascular Disorders; Peripheral Vascular Diseases; Coronary Disease; Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
To determine the incidence of type II diabetes and cardiovascular disease among Mexican-American and non-Hispanic whites in a 15 to 24 year follow-up of the San Antonio Heart Study 1 participants. Also, to perform a 15 to 24 year mortality follow-up of the cohort and to examine the "Hispanic paradox".

DETAILED DESCRIPTION:
BACKGROUND:

The San Antonio Heart Study 1 was a population-based survey of diabetes and cardiovascular risk factors in Mexican Americans and non-Hispanic whites conducted from 1979 to 1982. Participants included all men and non-pregnant women ages 24 to 64, who resided in households randomly sampled from three socio-culturally distinct neighborhoods of San Antonio. The low-income barrio residents were almost exclusively traditional Mexican-Americans. The middle-income neighborhood was ethnically balanced with equal numbers of Mexican Americans and Anglos whereas the upper income suburb was approximately 90 percent Anglo. Risk factors measured included obesity, glucose intolerance, hypertriglyceridemia, low levels of high density lipoprotein cholesterol, and blood pressure. The total number of people who were examined medically was 2,386, divided as follows: 1,288 Mexican Americans; 929 Anglos; and 169 other Hispanics such as Cubans. The San Antonio Heart Study 1 was designed to test the hypothesis that as Mexican Americans became progressively more affluent and accultured to mainstream United States culture, they would gradually lose their diabetic pattern of cardiovascular risk factors of obesity, diabetes, and hypertriglyceridemia.

Mexican Americans are the second largest minority group in the United States. Despite this, as recently as 1977, little was known about their health status. In recent years this situation has begun to change with publication of results from several major studies including the San Antonio Heart Study, the Starr County Study, and most recently the Hispanic Health and Nutrition Examination Survey (HHANES).

DESIGN NARRATIVE:

Beginning in 1987, each participant in the prospective San Antonio Heart Study 1 was recalled as close as possible to the eighth anniversary of his or her baseline examination and re-examined. Subjects had fasting lipid and lipoprotein determinations, a glucose tolerance test to diagnose incident cases of non-insulin dependent diabetes mellitus according to the National Diabetes Data Group criteria, blood pressure measurements, a resting electrocardiogram, and completed a questionnaire to elicit information on possible cardiovascular endpoints. Medical records were obtained to document the endpoints. Subjects with a history of peripheral vascular disease or diabetes had ankle/arm blood pressure ratios determined before and after exercise. Deaths were ascertained in the course of routine follow-up supplemented by search of state health department and National Death Index records. Death certificates were requested and for those certificates indicating diabetes or cardiovascular disease as the cause of death, hospital or physician records were requested and reviewed. Standardized criteria were used to validate cause of death. Endpoints included diabetes, sudden cardiac death, non-fatal (including silent) myocardial infarction, angina pectoris, cerebrovascular and peripheral vascular disease. The study was renewed in 1992 to continue follow-up.

The study was renewed in 1998 to perform a 15 to 24 year mortality follow-up of the cohort. Time dependencies in the ethnic mortality ratio were examined as well as other covariates such as biochemical parameters, hemodynamic variables, and anthropometric variables such as socioeconomic status, health care access and utilization and migrant status. A sample of 200 Mexican-American and 200 non-Hispanic white death certificates were verified by medical record review. The purpose of the review was to determine whether Mexican Americans, deemed to have died of cardiovascular causes based on medical record review, were more or less likely to have cardiovascular codes (ICDA 390-459) listed on their death certificates than non-Hispanic whites deemed to have died of these causes. The review aided in the interpretation of data relating to possible ethnic differences in cause-specific mortality based on death certificate coding.

The study should help to explain whether the "Hispanic paradox" is an artifact of underascertainment of deaths in this group. The "Hispanic paradox" refers to the concept that all-cause and cardiovascular (CV) mortality are widely thought to be lower in Hispanics, including Mexican Americans, than in non-Hispanic whites in the United States. Preliminary mortality data from this study suggest that all-cause mortality is actually higher in Mexican Americans than in non-Hispanic whites in San Antonio.

ELIGIBILITY:
No eligibility criteria

Ages: 24 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 1987-08; Study Completion 2003-07

CONTACTS AND LOCATIONS:
Overall Officials: Michael Stern, Principal Investigator — University of Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haffner SM, Mykkanen L, Gruber KK, Rainwater DL, Laakso M. Lack of association between sex hormones and Lp(a) concentrations in American and Finnish men. Arterioscler Thromb. 1994 Jan;14(1):19-24. doi: 10.1161/01.atv.14.1.19. PMID 8274474
- [Background] Haffner SM, Gonzales C, Valdez RA, Mykkanen L, Hazuda HP, Mitchell BD, Monterrosa A, Stern MP. Is microalbuminuria part of the prediabetic state? The Mexico City Diabetes Study. Diabetologia. 1993 Oct;36(10):1002-6. doi: 10.1007/BF02374491. PMID 8243847
- [Background] Haffner SM, Diehl AK, Valdez R, Mitchell BD, Hazuda HP, Morales P, Stern MP. Clinical gallbladder disease in NIDDM subjects. Relationship to duration of diabetes and severity of glycemia. Diabetes Care. 1993 Sep;16(9):1276-84. doi: 10.2337/diacare.16.9.1276. PMID 8404432
- [Background] Stern MP, Valdez RA, Haffner SM, Mitchell BD, Hazuda HP. Stability over time of modern diagnostic criteria for type II diabetes. Diabetes Care. 1993 Jul;16(7):978-83. doi: 10.2337/diacare.16.7.978. PMID 8359106
- [Background] Haffner SM, Mykkanen L, Stern MP, Valdez RA, Heisserman JA, Bowsher RR. Relationship of proinsulin and insulin to cardiovascular risk factors in nondiabetic subjects. Diabetes. 1993 Sep;42(9):1297-302. doi: 10.2337/diab.42.9.1297. PMID 8349041
- [Background] Stern MP, Morales PA, Valdez RA, Monterrosa A, Haffner SM, Mitchell BD, Hazuda HP. Predicting diabetes. Moving beyond impaired glucose tolerance. Diabetes. 1993 May;42(5):706-14. doi: 10.2337/diab.42.5.706. PMID 8482427
- [Background] Haffner SM, Morales PA, Gruber MK, Hazuda HP, Stern MP. Cardiovascular risk factors in non-insulin-dependent diabetic subjects with microalbuminuria. Arterioscler Thromb. 1993 Feb;13(2):205-10. doi: 10.1161/01.atv.13.2.205. PMID 8427856
- [Background] Morales PA, Mitchell BD, Valdez RA, Hazuda HP, Stern MP, Haffner SM. Incidence of NIDDM and impaired glucose tolerance in hypertensive subjects. The San Antonio Heart Study. Diabetes. 1993 Jan;42(1):154-61. doi: 10.2337/diab.42.1.154. PMID 8420812
- [Background] Haffner SM, Morales PA, Hazuda HP, Stern MP. Level of control of hypertension in Mexican Americans and non-Hispanic whites. Hypertension. 1993 Jan;21(1):83-8. doi: 10.1161/01.hyp.21.1.83. PMID 8418027
- [Background] Haffner SM, Miettinen H, Stern MP. Relatively more atherogenic coronary heart disease risk factors in prediabetic women than in prediabetic men. Diabetologia. 1997 Jun;40(6):711-7. doi: 10.1007/s001250050738. PMID 9222652
- [Background] Haffner SM, Miettinen H, Stern MP. Are risk factors for conversion to NIDDM similar in high and low risk populations? Diabetologia. 1997 Jan;40(1):62-6. doi: 10.1007/s001250050643. PMID 9028719
- [Background] Wei M, Stern MP, Haffner SM. Serum leptin levels in Mexican Americans and non-Hispanic whites: association with body mass index and cigarette smoking. Ann Epidemiol. 1997 Feb;7(2):81-6. doi: 10.1016/s1047-2797(96)00114-7. PMID 9099395
- [Background] Wei M, Gaskill SP, Haffner SM, Stern MP. Waist circumference as the best predictor of noninsulin dependent diabetes mellitus (NIDDM) compared to body mass index, waist/hip ratio and other anthropometric measurements in Mexican Americans--a 7-year prospective study. Obes Res. 1997 Jan;5(1):16-23. doi: 10.1002/j.1550-8528.1997.tb00278.x. PMID 9061711
- [Background] Haffner SM, Miettinen H, Gaskill SP, Stern MP. Decreased insulin action and insulin secretion predict the development of impaired glucose tolerance. Diabetologia. 1996 Oct;39(10):1201-7. doi: 10.1007/BF02658507. PMID 8897008
- [Background] Wei M, Valdez RA, Mitchell BD, Haffner SM, Stern MP, Hazuda HP. Migration status, socioeconomic status, and mortality rates in Mexican Americans and non-Hispanic whites: the San Antonio Heart Study. Ann Epidemiol. 1996 Jul;6(4):307-13. doi: 10.1016/s1047-2797(96)00026-9. PMID 8876841
- [Background] Haffner SM, Gingerich RL, Miettinen H, Stern MP. Leptin concentrations in relation to overall adiposity and regional body fat distribution in Mexican Americans. Int J Obes Relat Metab Disord. 1996 Oct;20(10):904-8. PMID 8910093
- [Background] Wei M, Mitchell BD, Haffner SM, Stern MP. Effects of cigarette smoking, diabetes, high cholesterol, and hypertension on all-cause mortality and cardiovascular disease mortality in Mexican Americans. The San Antonio Heart Study. Am J Epidemiol. 1996 Dec 1;144(11):1058-65. doi: 10.1093/oxfordjournals.aje.a008878. PMID 8942437
- [Background] Wei M, Gonzalez C, Haffner SM, O'Leary DH, Stern MP. Ultrasonographically assessed maximum carotid artery wall thickness in Mexico City residents and Mexican Americans living in San Antonio, Texas. Association with diabetes and cardiovascular risk factors. Arterioscler Thromb Vasc Biol. 1996 Nov;16(11):1388-92. doi: 10.1161/01.atv.16.11.1388. PMID 8911278
- [Background] Gonzalez Villalpando C, Stern MP, Arredondo Perez B, Martinez Diaz S, Islas Andrade S, Revilla C, Gonzalez Villalpando ME, Rivera Martinez D. Nephropathy in low income diabetics: the Mexico City Diabetes Study. Arch Med Res. 1996 Autumn;27(3):367-72. PMID 8854397
- [Background] Haffner SM, Miettinen H, Gaskill SP, Stern MP. Metabolic precursors of hypertension. The San Antonio Heart Study. Arch Intern Med. 1996 Sep 23;156(17):1994-2001. PMID 8823152
- [Background] Gonzalez Villalpando C, Stern MP, Arredondo Perez B, Martinez Diaz S, Haffner S. Undiagnosed hypercholesterolemia: a serious health challenge. The Mexico City Diabetes Study. Arch Med Res. 1996 Spring;27(1):19-23. PMID 8867362
- [Background] Haffner SM, Stern MP, Miettinen H, Robbins D, Howard BV. Apolipoprotein E polymorphism and LDL size in a biethnic population. Arterioscler Thromb Vasc Biol. 1996 Sep;16(9):1184-8. doi: 10.1161/01.atv.16.9.1184. PMID 8792773
- [Background] Haffner SM, Miettinen H, Stern MP. Nondiabetic Mexican-Americans do not have reduced insulin responses relative to nondiabetic non-Hispanic whites. Diabetes Care. 1996 Jan;19(1):67-9. doi: 10.2337/diacare.19.1.67. PMID 8720538
- [Background] Haffner SM, Miettinen H, Stern MP, Agil A, Jialal I. Plasma oxidizability in Mexican-Americans and non-Hispanic whites. Metabolism. 1996 Jul;45(7):876-81. doi: 10.1016/s0026-0495(96)90163-8. PMID 8692025
- [Background] Haffner SM, Stern MP, Miettinen H, Wei M, Gingerich RL. Leptin concentrations in diabetic and nondiabetic Mexican-Americans. Diabetes. 1996 Jun;45(6):822-4. doi: 10.2337/diab.45.6.822. PMID 8635660
- [Background] Haffner SM, Miettinen H, Stern MP. Insulin secretion and resistance in nondiabetic Mexican Americans and non-Hispanic whites with a parental history of diabetes. J Clin Endocrinol Metab. 1996 May;81(5):1846-51. doi: 10.1210/jcem.81.5.8626845.
- [Background] Haffner SM, Agil A, Mykkanen L, Stern MP, Jialal I. Plasma oxidizability in subjects with normal glucose tolerance, impaired glucose tolerance, and NIDDM. Diabetes Care. 1995 May;18(5):646-53. doi: 10.2337/diacare.18.5.646. PMID 8586002
- [Background] Haffner SM, Mykkanen L, Robbins D, Valdez R, Miettinen H, Howard BV, Stern MP, Bowsher R. A preponderance of small dense LDL is associated with specific insulin, proinsulin and the components of the insulin resistance syndrome in non-diabetic subjects. Diabetologia. 1995 Nov;38(11):1328-36. doi: 10.1007/BF00401766. PMID 8582543
- [Background] Valdez R, Gonzalez-Villalpando C, Mitchell BD, Haffner SM, Stern MP. Differential impact of obesity in related populations. Obes Res. 1995 Sep;3 Suppl 2:223s-232s. doi: 10.1002/j.1550-8528.1995.tb00468.x. PMID 8581781
- [Background] Monterrosa AE, Haffner SM, Stern MP, Hazuda HP. Sex difference in lifestyle factors predictive of diabetes in Mexican-Americans. Diabetes Care. 1995 Apr;18(4):448-56. doi: 10.2337/diacare.18.4.448. PMID 7497852
- [Background] Haffner SM, Miettinen H, Gaskill SP, Stern MP. Decreased insulin secretion and increased insulin resistance are independently related to the 7-year risk of NIDDM in Mexican-Americans. Diabetes. 1995 Dec;44(12):1386-91. doi: 10.2337/diab.44.12.1386. PMID 7589843
- [Background] Haffner SM, Stern MP, Miettinen H, Gingerich R, Bowsher RR. Higher proinsulin and specific insulin are both associated with a parental history of diabetes in nondiabetic Mexican-American subjects. Diabetes. 1995 Oct;44(10):1156-60. doi: 10.2337/diab.44.10.1156. PMID 7556950
- [Background] Valdez R, Howard BV, Stern MP, Haffner SM. Apolipoprotein E polymorphism and insulin levels in a biethnic population. Diabetes Care. 1995 Jul;18(7):992-1000. doi: 10.2337/diacare.18.7.992. PMID 7555562
- [Background] Mitchell BD, Gonzalez Villalpando C, Arredondo Perez B, Garcia MS, Valdez R, Stern MP. Myocardial infarction and cardiovascular risk factors in Mexico City and San Antonio, Texas. Arterioscler Thromb Vasc Biol. 1995 Jun;15(6):721-5. doi: 10.1161/01.atv.15.6.721. PMID 7773724
- [Background] Haffner SM, Stern MP, Mitchell BD, Hazuda HP, Patterson JK. Incidence of type II diabetes in Mexican Americans predicted by fasting insulin and glucose levels, obesity, and body-fat distribution. Diabetes. 1990 Mar;39(3):283-8. doi: 10.2337/diab.39.3.283. PMID 2407581
- [Background] Haffner SM, Stern MP, Hazuda HP, Mitchell BD, Patterson JK. Cardiovascular risk factors in confirmed prediabetic individuals. Does the clock for coronary heart disease start ticking before the onset of clinical diabetes? JAMA. 1990 Jun 6;263(21):2893-8. doi: 10.1001/jama.263.21.2893. PMID 2338751
- [Background] Haffner SM, Stern MP, Gruber MK, Hazuda HP, Mitchell BD, Patterson JK. Microalbuminuria. Potential marker for increased cardiovascular risk factors in nondiabetic subjects? Arteriosclerosis. 1990 Sep-Oct;10(5):727-31. doi: 10.1161/01.atv.10.5.727. PMID 2403300
- [Background] Mitchell BD, Hazuda HP, Haffner SM, Patterson JK, Stern MP. Myocardial infarction in Mexican-Americans and non-Hispanic whites. The San Antonio Heart Study. Circulation. 1991 Jan;83(1):45-51. doi: 10.1161/01.cir.83.1.45. PMID 1984897
- [Background] Haffner SM, Mitchell BD, Stern MP, Hazuda HP, Patterson JK. Public health significance of upper body adiposity for non-insulin dependent diabetes mellitus in Mexican Americans. Int J Obes Relat Metab Disord. 1992 Mar;16(3):177-84. PMID 1317826
- [Background] Gonzalez-Villalpando C, Stern MP, Villalpando E, Hazuda H, Haffner SM, Lisci E. [Prevalence of diabetes and glucose intolerance in a urban population at a low economic level]. Rev Invest Clin. 1992 Jul-Sep;44(3):321-8. Spanish. PMID 1488576
- [Background] Pugh JA, Tuley MR, Hazuda HP, Stern MP. The influence of outpatient insurance coverage on the microvascular complications of non-insulin-dependent diabetes in Mexican Americans. J Diabetes Complications. 1992 Oct-Dec;6(4):236-41. doi: 10.1016/1056-8727(92)90058-s. PMID 1482781
- [Background] Haffner SM, Gruber KK, Aldrete G Jr, Morales PA, Stern MP, Tuttle KR. Increased lipoprotein(a) concentrations in chronic renal failure. J Am Soc Nephrol. 1992 Nov;3(5):1156-62. doi: 10.1681/ASN.V351156. PMID 1482754
- [Background] Haffner SM, Gruber KK, Morales PA, Hazuda HP, Valdez RA, Mitchell BD, Stern MP. Lipoprotein(a) concentrations in Mexican Americans and non-Hispanic whites: the San Antonio Heart Study. Am J Epidemiol. 1992 Nov 1;136(9):1060-8. doi: 10.1093/oxfordjournals.aje.a116571. PMID 1462966
- [Background] Stern MP, Morales PA, Haffner SM, Valdez RA. Hyperdynamic circulation and the insulin resistance syndrome ("syndrome X"). Hypertension. 1992 Dec;20(6):802-8. doi: 10.1161/01.hyp.20.6.802. PMID 1452296
- [Background] Haffner SM, Morales PA, Stern MP, Gruber MK. Lp(a) concentrations in NIDDM. Diabetes. 1992 Oct;41(10):1267-72. doi: 10.2337/diab.41.10.1267. PMID 1397699
- [Background] Haffner SM, Tuttle KR, Rainwater DL. Lack of change of lipoprotein (a) concentration with improved glycemic control in subjects with type II diabetes. Metabolism. 1992 Feb;41(2):116-20. doi: 10.1016/0026-0495(92)90136-x. PMID 1531244
- [Background] Stern MP, Mitchell BD, Haffner SM, Hazuda HP. Does glycemic control of type II diabetes suffice to control diabetic dyslipidemia? A community perspective. Diabetes Care. 1992 May;15(5):638-44. doi: 10.2337/diacare.15.5.638. PMID 1516483
- [Background] Haffner SM, Ferrannini E, Hazuda HP, Stern MP. Clustering of cardiovascular risk factors in confirmed prehypertensive individuals. Hypertension. 1992 Jul;20(1):38-45. doi: 10.1161/01.hyp.20.1.38. PMID 1618551
- [Background] Haffner SM, Valdez RA, Hazuda HP, Mitchell BD, Morales PA, Stern MP. Prospective analysis of the insulin-resistance syndrome (syndrome X). Diabetes. 1992 Jun;41(6):715-22. doi: 10.2337/diab.41.6.715. PMID 1587398
- [Background] Haffner SM, Stern MP, Watanabe RM, Bergman RN. Relationship of insulin clearance and secretion to insulin sensitivity in non-diabetic Mexican Americans. Eur J Clin Invest. 1992 Mar;22(3):147-53. doi: 10.1111/j.1365-2362.1992.tb01819.x. PMID 1582438
- [Background] Haffner SM, Mitchell BD, Valdez RA, Hazuda HP, Morales PA, Stern MP. Eight-year incidence of hypertension in Mexican-Americans and non-Hispanic whites. The San Antonio Heart Study. Am J Hypertens. 1992 Mar;5(3):147-53. doi: 10.1093/ajh/5.3.147. PMID 1575941
- [Background] Jameel N, Pugh JA, Mitchell BD, Stern MP. Dietary protein intake is not correlated with clinical proteinuria in NIDDM. Diabetes Care. 1992 Feb;15(2):178-83. doi: 10.2337/diacare.15.2.178. PMID 1547674
- [Background] Haffner SM, Dunn JF, Katz MS. Relationship of sex hormone-binding globulin to lipid, lipoprotein, glucose, and insulin concentrations in postmenopausal women. Metabolism. 1992 Mar;41(3):278-84. doi: 10.1016/0026-0495(92)90271-b. PMID 1542267
- [Background] Stern MP. Kelly West Lecture. Primary prevention of type II diabetes mellitus. Diabetes Care. 1991 May;14(5):399-410. doi: 10.2337/diacare.14.5.399. PMID 2060452
- [Background] Haffner SM, Hazuda HP, Mitchell BD, Patterson JK, Stern MP. Increased incidence of type II diabetes mellitus in Mexican Americans. Diabetes Care. 1991 Feb;14(2):102-8. doi: 10.2337/diacare.14.2.102. PMID 2060411
- [Background] Hazuda HP, Mitchell BD, Haffner SM, Stern MP. Obesity in Mexican American subgroups: findings from the San Antonio Heart Study. Am J Clin Nutr. 1991 Jun;53(6 Suppl):1529S-1534S. doi: 10.1093/ajcn/53.6.1529S. PMID 2031483
- [Background] Stern MP, Patterson JK, Mitchell BD, Haffner SM, Hazuda HP. Overweight and mortality in Mexican Americans. Int J Obes. 1990 Jul;14(7):623-9. PMID 2228397
- [Background] Haffner SM, Gonzalez C, Miettinen H, Howard BV, Stern MP. LDL size and subclass pattern in Mexico City residents and San Antonio Mexican Americans. Arterioscler Thromb Vasc Biol. 1995 Dec;15(12):2136-41. doi: 10.1161/01.atv.15.12.2136. PMID 7489234
- [Background] Haffner SM, Karhapaa P, Rainwater DL, Mykkanen L, Aldrete G Jr, Laakso M. Insulin sensitivity and Lp(a) concentrations in normoglycemic men. Diabetes Care. 1995 Feb;18(2):193-9. doi: 10.2337/diacare.18.2.193. PMID 7729297
- [Background] Haffner SM, Mykkanen L, Valdez RA, Stern MP, Holloway DL, Monterrosa A, Bowsher RR. Disproportionately increased proinsulin levels are associated with the insulin resistance syndrome. J Clin Endocrinol Metab. 1994 Dec;79(6):1806-10. doi: 10.1210/jcem.79.6.7989488.
- [Background] Haffner S, Gonzalez Villalpando C, Hazuda HP, Valdez R, Mykkanen L, Stern M. Prevalence of hypertension in Mexico City and San Antonio, Texas. Circulation. 1994 Sep;90(3):1542-9. doi: 10.1161/01.cir.90.3.1542. PMID 8087960
- [Background] Gonzelez C, Stern MP, Mitchell BD, Valdez RA, Haffner SM, Perez BA. Clinical characteristics of type II diabetic subjects consuming high versus low carbohydrate diets in Mexico City and San Antonio, Texas. Diabetes Care. 1994 May;17(5):397-404. doi: 10.2337/diacare.17.5.397. PMID 8062606
- [Background] Stern MP, Wei M. Do Mexican Americans really have low rates of cardiovascular disease? Prev Med. 1999 Dec;29(6 Pt 2):S90-5. doi: 10.1006/pmed.1998.0464. PMID 10641824
- [Background] Gonzalez-Villalpando C, Gonzalez-Villalpando ME, Rivera Martinez D, Stern MP. [Incidence and progression of diabetic retinopathy in low income population of Mexico City]. Rev Invest Clin. 1999 May-Jun;51(3):141-50. Spanish. PMID 10466004
- [Background] Gonzalez-Villalpando C, Stern MP, Haffner SM, Gonzalez Villapando ME, Gaskill S, Rivera Martinez D. Prevalence of hypertension in a Mexican population according to the Sixth Report of the Joint National Committee on Prevention, Detection, Evaluation and Treatment of High Blood Pressure. J Cardiovasc Risk. 1999 Jun;6(3):177-81. doi: 10.1177/204748739900600309. PMID 10463145
- [Background] Haffner SM, Miettinen H, Mykkanen L, Stern MP. Leptin concentrations are associated with higher proinsulin and insulin concentrations but a lower proinsulin/insulin ratio in non-diabetic subjects. Int J Obes Relat Metab Disord. 1998 Sep;22(9):899-905. doi: 10.1038/sj.ijo.0800679. PMID 9756249
- [Background] Wei M, Gibbons LW, Mitchell TL, Kampert JB, Stern MP, Blair SN. Low fasting plasma glucose level as a predictor of cardiovascular disease and all-cause mortality. Circulation. 2000 May 2;101(17):2047-52. doi: 10.1161/01.cir.101.17.2047. PMID 10790345
- [Background] Haffner SM, Mykkanen L, Festa A, Burke JP, Stern MP. Insulin-resistant prediabetic subjects have more atherogenic risk factors than insulin-sensitive prediabetic subjects: implications for preventing coronary heart disease during the prediabetic state. Circulation. 2000 Mar 7;101(9):975-80. doi: 10.1161/01.cir.101.9.975. PMID 10704163
- [Background] Lorenzo C, Serrano-Rios M, Martinez-Larrad MT, Gabriel R, Williams K, Gonzalez-Villalpando C, Stern MP, Hazuda HP, Haffner S. Prevalence of hypertension in Hispanic and non-Hispanic white populations. Hypertension. 2002 Feb;39(2):203-8. doi: 10.1161/hy0202.103439. PMID 11847184
- [Background] del Rincon ID, Williams K, Stern MP, Freeman GL, Escalante A. High incidence of cardiovascular events in a rheumatoid arthritis cohort not explained by traditional cardiac risk factors. Arthritis Rheum. 2001 Dec;44(12):2737-45. doi: 10.1002/1529-0131(200112)44:123.0.CO;2-%23. PMID 11762933
- [Background] Lorenzo C, Serrano-Rios M, Martinez-Larrad MT, Gabriel R, Williams K, Gonzalez-Villalpando C, Stern MP, Hazuda HP, Haffner SM. Was the historic contribution of Spain to the Mexican gene pool partially responsible for the higher prevalence of type 2 diabetes in mexican-origin populations? The Spanish Insulin Resistance Study Group, the San Antonio Heart Study, and the Mexico City Diabetes Study. Diabetes Care. 2001 Dec;24(12):2059-64. doi: 10.2337/diacare.24.12.2059. PMID 11723083
- [Background] Burke JP, Williams K, Haffner SM, Villalpando CG, Stern MP. Elevated incidence of type 2 diabetes in San Antonio, Texas, compared with that of Mexico City, Mexico. Diabetes Care. 2001 Sep;24(9):1573-8. doi: 10.2337/diacare.24.9.1573. PMID 11522701
- [Background] Burke JP, Hazuda HP, Stern MP. Rising trend in obesity in Mexican Americans and non-Hispanic whites: is it due to cigarette smoking cessation? Int J Obes Relat Metab Disord. 2000 Dec;24(12):1689-94. doi: 10.1038/sj.ijo.0801439. PMID 11126225
- [Background] Stern MP, Williams K, Haffner SM. Identification of persons at high risk for type 2 diabetes mellitus: do we need the oral glucose tolerance test? Ann Intern Med. 2002 Apr 16;136(8):575-81. doi: 10.7326/0003-4819-136-8-200204160-00006. PMID 11955025
- [Background] Stern MP, Fatehi P, Williams K, Haffner SM. Predicting future cardiovascular disease: do we need the oral glucose tolerance test? Diabetes Care. 2002 Oct;25(10):1851-6. doi: 10.2337/diacare.25.10.1851. PMID 12351490
- [Background] Hunt KJ, Williams K, Resendez RG, Hazuda HP, Haffner SM, Stern MP. All-cause and cardiovascular mortality among diabetic participants in the San Antonio Heart Study: evidence against the "Hispanic Paradox". Diabetes Care. 2002 Sep;25(9):1557-63. doi: 10.2337/diacare.25.9.1557. PMID 12196427
- [Background] Lorenzo C, Serrano-Rios M, Martinez-Larrad MT, Gabriel R, Williams K, Gomez-Gerique JA, Stern MP, Haffner SM. Central adiposity determines prevalence differences of the metabolic syndrome. Obes Res. 2003 Dec;11(12):1480-7. doi: 10.1038/oby.2003.198. PMID 14694212
- [Background] Ferrannini E, Nannipieri M, Williams K, Gonzales C, Haffner SM, Stern MP. Mode of onset of type 2 diabetes from normal or impaired glucose tolerance. Diabetes. 2004 Jan;53(1):160-5. doi: 10.2337/diabetes.53.1.160. PMID 14693710
- [Background] Hunt KJ, Resendez RG, Williams K, Haffner SM, Stern MP, Hazuda HP. All-cause and cardiovascular mortality among Mexican-American and non-Hispanic White older participants in the San Antonio Heart Study- evidence against the "Hispanic paradox". Am J Epidemiol. 2003 Dec 1;158(11):1048-57. doi: 10.1093/aje/kwg249. PMID 14630600
- [Background] Del Rincon I, Williams K, Stern MP, Freeman GL, O'Leary DH, Escalante A. Association between carotid atherosclerosis and markers of inflammation in rheumatoid arthritis patients and healthy subjects. Arthritis Rheum. 2003 Jul;48(7):1833-40. doi: 10.1002/art.11078. PMID 12847676
- [Background] Lorenzo C, Okoloise M, Williams K, Stern MP, Haffner SM; San Antonio Heart Study. The metabolic syndrome as predictor of type 2 diabetes: the San Antonio heart study. Diabetes Care. 2003 Nov;26(11):3153-9. doi: 10.2337/diacare.26.11.3153. PMID 14578254
- [Background] Burke JP, Williams K, Narayan KM, Leibson C, Haffner SM, Stern MP. A population perspective on diabetes prevention: whom should we target for preventing weight gain? Diabetes Care. 2003 Jul;26(7):1999-2004. doi: 10.2337/diacare.26.7.1999. PMID 12832302
- [Background] Hanley AJ, Williams K, Gonzalez C, D'Agostino RB Jr, Wagenknecht LE, Stern MP, Haffner SM; San Antonio Heart Study; Mexico City Diabetes Study; Insulin Resistance Atherosclerosis Study. Prediction of type 2 diabetes using simple measures of insulin resistance: combined results from the San Antonio Heart Study, the Mexico City Diabetes Study, and the Insulin Resistance Atherosclerosis Study. Diabetes. 2003 Feb;52(2):463-9. doi: 10.2337/diabetes.52.2.463. PMID 12540622
- [Background] Meigs JB, Williams K, Sullivan LM, Hunt KJ, Haffner SM, Stern MP, Gonzalez Villalpando C, Perhanidis JS, Nathan DM, D'Agostino RB Jr, D'Agostino RB Sr, Wilson PW. Using metabolic syndrome traits for efficient detection of impaired glucose tolerance. Diabetes Care. 2004 Jun;27(6):1417-26. doi: 10.2337/diacare.27.6.1417. PMID 15161798
- [Background] Stern MP, Williams K, Gonzalez-Villalpando C, Hunt KJ, Haffner SM. Does the metabolic syndrome improve identification of individuals at risk of type 2 diabetes and/or cardiovascular disease? Diabetes Care. 2004 Nov;27(11):2676-81. doi: 10.2337/diacare.27.11.2676. PMID 15505004
- [Background] Hunt KJ, Resendez RG, Williams K, Haffner SM, Stern MP; San Antonio Heart Study. National Cholesterol Education Program versus World Health Organization metabolic syndrome in relation to all-cause and cardiovascular mortality in the San Antonio Heart Study. Circulation. 2004 Sep 7;110(10):1251-7. doi: 10.1161/01.CIR.0000140762.04598.F9. Epub 2004 Aug 23. PMID 15326061